CLINICAL TRIAL: NCT01736657
Title: Evaluation of the Spectra Optia Apheresis Red Blood Cell Exchange Protocol in Patients With Sickle Cell Disease.
Brief Title: Evaluation of Spectra Optia Red Blood Cell Exchange in Sickle Cell Patients
Acronym: ESSENTIAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Terumo BCT (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTS-5001
Record Dates: First submitted 2012-11-27; First posted 2012-11-29 (Estimated); Results first posted 2014-07-14 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2014-01

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Red cell exchange in sickle cell (Experimental): Open arm; Red cell blood exchange for patients with sickle cell disease
  Interventions: Device: Red blood cell exchange in sickle cell

INTERVENTIONS:
Device: Red blood cell exchange in sickle cell — One Red Blood Cell Exchange using Spectra Optia Apheresis System per enrolled patient
  Other Names: Specta Optia Apheresis System

SUMMARY:
The purpose of this study is to evaluate the performance of the Spectra Optia system red blood cell exchange (RBCx) protocols (exchange and depletion/exchange) in study participants with sickle cell disease.

DETAILED DESCRIPTION:
Evaluate the performance of the Spectra Optia system red blood cell exchange (RBCx) protocols (exchange and depletion/exchange) in study participants with sickle cell disease. Open label design.

ELIGIBILITY:
Inclusion Criteria:

* At least 12 years old
* Enrolled in a program of regular red blood cell exchange (RBCx) to prevent symptoms/complications of sickle cell disease (SCD) or Initiating a program of regular RBCx or Receiving RBCx as a pre-surgical procedure.
* Medically stable
* Previous documentation of diagnosis by hemoglobin electrophoresis of a type of sickle cell disorder requiring RBCx.
* Sufficient vascular access to accommodate the RBCx procedure as determined by the apheresis technician performing the procedure or phlebotomist responsible for obtaining intravenous access.
* Availability of sickle trait negative, leukoreduced, ABO blood group, Rhesus factor D (Rh (D)) compatible, unexpired replacement blood. See Glossary for definition of replacement blood.
* Able to commit to the study follow-up schedule.
* Agree to report adverse events (AEs) during the required reporting period.

Exclusion Criteria:

* Inability to obtain informed consent/assent from patient, or permission from parent or guardian.
* Pregnancy (negative serum pregnancy test required for females of childbearing potential).
* Life expectancy is fewer than 30 days from time of procedure.
* Incarcerated or a ward of the court.
* Refusal of blood products.
* Failure to comply with site standard requirements for cessation of medications (e.g., angiotensin converting enzyme (ACE) inhibitors) that interfere with or increase risk of RBCx procedures.
* History of drug or alcohol abuse that, in the opinion of the investigator, could affect the ability of the patient to comply with the study requirements Inability to comply with the protocol in the opinion of the investigator.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2012-11; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keith Quirolo, MD, Principal Investigator — Children's Hospital and Research Center at Oakland
Locations (5):
- United States (5):
  - Children's of Alabama, Birmingham, Alabama
  - Children's Hospital and Research Center at Oakland, Oakland, California
  - University of Colorado at Denver, Aurora, Colorado
  - Kosair Children's Hospital, Louisville, Kentucky
  - Johns Hopkins Medical, Baltimore, Maryland

REFERENCES:
- [Derived] Quirolo K, Bertolone S, Hassell K, Howard T, King KE, Rhodes DK, Bill J. The evaluation of a new apheresis device for automated red blood cell exchange procedures in patients with sickle cell disease. Transfusion. 2015 Apr;55(4):775-81. doi: 10.1111/trf.12891. Epub 2014 Oct 21. PMID 25330984

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: Nov 2012 through May 2013
Pre-assignment Details: Evaluable population includes 60 pts. Terumo Optia Trainer was present for Optia Operator support for 12 procedures, called "lead-in" procedures: these were not included in efficacy analysis, but were included in safety analysis (full analysis set).
Groups:
- Red Blood Cell Exchange for Patients With Sickle Cell Disease: Red blood cell exchange or depletion/exchange for patients with sickle cell disease : The purpose of this study is to evaluate the performance of the Red Blood Cell Exchange protocol on the Spectra Optia Apheresis System.
Period: Overall Study
Arm/Group | Red Blood Cell Exchange for Patients With Sickle Cell Disease
Started | 73
Completed | 72
Not Completed | 1
Not completed — insufficient vascular access | 1

BASELINE CHARACTERISTICS:
Population: Seventy-two patients were in safety analysis and 60 patients (evaluable popluation) were analyzed in the efficacy analysis. The 12 patients not in the efficacy analysis were "lead-in" patients and the RBCX procedures were conducted as the last phase in Operator training on the device.
Arm/Group | Red Blood Cell Exchange for Patients With Sickle Cell Disease
Number analyzed (Participants) | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 26
  Between 18 and 65 years | 46
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.0 (10.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 43
Region of Enrollment [Number; unit: participants]
  United States | 72

OUTCOME MEASURES:

1. Primary Outcome: Mean Ratio Actual Fraction of Cells Remaining (FCRa; as Measured by Post-Procedure % HbS) to the Predicted Fraction of Cells Remaining (FCRp; as Predicted by the Spectra Optia System FCR Algorithm Multiplied by the Pre-Procedure % HbS)
Description: The primary endpoint evaluated the mean ratio of the Actual Fraction of Cells Remaining (FCRa: as measured by Post-Procedure % HbS) to the Predicted Fraction of Cells Remaining (FCRp: as predicted by the Spectra Optia system FCR algorithm multiplied by the Pre-Procedure % HbS), in the evaluable population (60 pts). The pre-defined range for the mean ratio of the FCRa to the FCRp was 0.75 to 1.25.
Time Frame: Length of the procedure
Population: 60 patients analyzed, 73 enrolled:12 patients were lead-in patients whereby Optia Operators completed their training and data from those procedures were not included in the efficacy analysis (60 pts), but were included in the safety analysis (72 patients); 1 patient was consented but withdrawn prior to procedure due to lack of vascular access.
Measure: Mean (95% Confidence Interval); unit: ratio
Arm/Group | Red Blood Cell Exchange for Patients With Sickle Cell Disease
Number analyzed (Participants) | 60
ratio | 0.9 [0.855 to 0.941]

2. Secondary Outcome: Procedural Success of the Spectra Optia System in the Evaluable Population
Description: The procedural success of the Spectra Optia System is defined as the ability of the device to complete a red blood cell exchange (RBCx) and to obtain a satisfactory exchange by lowering the patient's hemoglobin S, as determined by the investigator in the evaluable population (60 pts).
Time Frame: Length of the procedure
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Red Blood Cell Exchange for Patients With Sickle Cell Disease
Number analyzed (Participants) | 60
percentage of participants | 100

3. Secondary Outcome: Spectra Optia System's Ability to Achieve the Desired Final Hematocrit in the Evaluable Population
Description: Measurement of the patient post-procedure hematocrit compared to the final target hematocrit calculated by the Spectra Optia Apheresis System. Final target hematocrit was calculated by tracking the number of red cells coming into the system versus the number of red cells removed.
Time Frame: Length of the procedure
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: ratio
Arm/Group | Red Blood Cell Exchange for Patients With Sickle Cell Disease
Number analyzed (Participants) | 60
ratio | 1.03 [1.011 to 1.045]

4. Secondary Outcome: Device-related Serious Adverse Events (SAE) in the Full Analysis Set
Description: Device-related serious adverse events (SAE) in the Full Analysis Set (72 patients).
Time Frame: upon signing consent to 24 hours post-procedure
Population: Seventy-three enrolled: 12 were lead-in patients whereby Optia Operators completed their training and data from those procedures were not included in the efficacy analysis (60 patients), but these patients were included in safety analysis as Full Analysis Set; 1 patient was consented but withdrawn prior to procedure due to lack of vascular access.
Measure: Number; unit: participants
Arm/Group | Red Blood Cell Exchange for Patients With Sickle Cell Disease
Number analyzed (Participants) | 72
participants | 0

ADVERSE EVENTS:
Arm/Group | Red Blood Cell Exchange for Patients With Sickle Cell Disease
Serious Adverse Events (participants affected / at risk) | 0/72
Other Adverse Events (participants affected / at risk) | 10/72
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Red Blood Cell Exchange for Patients With Sickle Cell Disease (N=72)
Nausea (Gastrointestinal disorders) | 4 (4)
Dizziness (Nervous system disorders) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If Study Site is performing services in a multi-center Study, it agrees not to independently publish, publicly disclose, present or discuss any results of or information pertaining to the Study until a multi-center manuscript is published; provided however, that if a multi-center manuscript is not published within one year after completion of the Study at all Study sites, Study Site may publish the Study data generated by Study Site